CLINICAL TRIAL: NCT05446519
Title: Descriptive Study of Anxiety and/or Depressive Disorders in a Population of Airline Pilots Employed in France and Unionized at the SNPL
Brief Title: Anxiety and / or Depressive Disorders in a Population of French Airline Pilot
Acronym: AEROPSY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22-PP-09
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Anxiety Disorders; Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — Survey is proposed to all pilots who are members of the National Union of Airline Pilots

SUMMARY:
Throughout their career, the medical abilities of airline pilots are regularly assessed. This population is exposed to occupational constraints and risks, in particular psychosocial, and could constitute a population at risk of developing anxiety and/or depressive disorders. However, mental health remains difficult to apprehend in this population because of a strong stigmatization of mental disorders and the risk of loss of medical certification to fly. In the literature, there are very few studies dealing with mental disorders in airline pilots and the results are heterogeneous, with a prevalence of anxiety and/or depressive disorders ranging from 1.9 to 12.6%. There is no study of this type among airline pilots employed in France. Therefore it seems useful to determine the prevalence of anxiety and/or depressive disorders in this population and to describe the co-factors associated with these disorders.

ELIGIBILITY:
Inclusion Criteria:

* Airline pilot, employed in France and unionized at the Syndicat National des Pilote de Ligne (SNPL)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Airline pilot, employed in France and unionized at the Syndicat National des Pilote de Ligne (SNPL)
Sampling Method: Non-Probability Sample
Enrollment: 870 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Depressive and anxiety disorders | at baseline
  Anxiety and depressive disorders as measured by Hospital Anxiety and Depression Scale (HAD-S). The HADS consists of 14 items, seven items indicating anxiety and seven items indicating depression. The answer format offers four options, scored with values from 0 to 3. This results in scale values between 0 and 21 for each scale. Three ranges were defined by the original test authors: 0-7 (non-cases), 8-10 (doubtful cases), and 11-21 (cases)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No